CLINICAL TRIAL: NCT06544382
Title: Rehabilitation and Return to Everyday Life for Patients With Long COVID
Status: Active, not recruiting | Type: Observational
Sponsor: Defactum, Central Denmark Region (Other Government)
Collaborators: Aarhus University Hospital (Other); VIA University College (Other); University of Aarhus (Other); Aarhus Municipality, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: Long COVID rehabilitation
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Long COVID
Keywords: Rehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Patients from Aarhus Municipality, Central Denmark Region, Denmark, receiving The Long COVID Rehabilitation Intervention.
  Interventions: Other: The Long COVID Rehabilitation Intervention
- Control group: Patients from the other municipalities of Central Denmark Region, Denmark, receiving a less structured rehabilitation programme with individual session and few group options with patients with long COVID or mixed diagnoses.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: The Long COVID Rehabilitation Intervention — The intervention is a structured rehabilitation intervention with a duration of minimum 3 months comprising 4-12 individual sessions and 1-4 group-based courses delivered by physiotherapists and occupational therapists.
  Groups: Intervention group
Other: Usual care — A less structured rehabilitation programme comprising individual session with a few group options with patients with long COVID or mixed diagnoses.
  Groups: Control group

SUMMARY:
This non-randomised controlled trial will investigate if patients with long COVID receiving a structured and group-based rehabilitation intervention (The Long COVID Rehabilitation Intervention) will report a difference in mean change in self-reported mental fatigue measured by Mental Fatigue Scale and will report a mean difference in weeks of sick-leave obtained through the Danish Register for Evaluation of Marginalisation compared to usual practise over a 12-month follow-up period. Alongside the effectiveness evaluation, a economic evaluation study and process evaluation study will be conducted,

Patients from Aarhus Municipality, Central Denmark Region, Denmark, receive The Long COVID Rehabilitation Intervention and will be allocated to the intervention group. Patients receiving rehabilitation in the other municipalities of Central Denmark Region, Denmark, will be allocated to the control group. Alongside this, a health economic study and a process evaluation study will be conducted.

DETAILED DESCRIPTION:
The study is a non-randomised controlled trial with 12-month follow-up. Alongside this, a health economic study and process evaluation study will be conducted in line with the British Medical Research Council's framework for development and evaluation of complex interventions. The study will be reported in three separate scientific papers for each evaluation study.

This study aims to evaluate the effectiveness of a structured and group-based rehabilitation intervention, called The Long COVID Rehabilitation Intervention, with the goal to optimise the rehabilitation of patients experiencing long-term symptoms after COVID-19 (long COVID).

The primary hypothesis: A structured and personalised rehabilitation intervention for patients with long COVID is more effective evaluated on sick leave, mental fatigue and disability compared to usual rehabilitation.

To evaluate the aim, the intervention group (patients receiving The Long COVID Rehabilitation Intervention in Aarhus Municipality, Central Denmark Region, Denmark) will be compared to a control group (patients receiving rehabilitation in the 18 other municipalities in Central Denmark Region, Denmark).

The data will be handled in accordance with the World Medical Association Coherence Declaration of Helsinki and with the General Data Protection Regulation. The study is approved by the Danish Regional Data Protection Agency (J.nr. 1-16-02-655-20).

The intervention group (patients from Aarhus Municipality, Central Denmark Region) received The Long COVID Rehabilitation Intervention; a rehabilitation programme with a duration of minimum 3 months comprising 4-12 individual sessions and 1-4 group-based courses with physiotherapists and occupational therapists. The control group (patients from the other 18 municipalities in Central Denmark region) received the rehabilitation interventions delivered in their home municipality which were generally less structured with more individual sessions compared to the intervention group. Based on a systematic identification through semi-structured interviews with representatives from all 19 municipalities in Central Denmark Region, the rehabilitation provided for long COVID patients was described for each municipality using the TIDieR template. Throughout the study period, it will be explored if it is possible to divide the control groups into two subgroups depending on the rehabilitation provided in the municipalities.

With a mean Mental Fatigue Scale score of 18.6 (SD: 5.6), a minimal clinical important difference of 2 points, a power of 80% and a two-sided significance level of 0.05, a total study population of 375 (125 patients in each group) patients should be included. To account for a 20% loss to follow-up, the total number is 450 patients. For long term sick leave, a power calculation will be performed during the fall 2024 based on data from an ongoing study.

Data are collected through questionnaires sent out electronically and through register data. Sociodemographic characteristics (sex, age, and self-reported living status, education, work status and occupation) and self-reported information on main symptoms and time since infection is collected at inclusion. Study data are collected and managed using REDCap electronic data capture tools.

Descriptive statistics will be conducted to describe sociodemographic characteristics. To evaluate the effectiveness of the intervention, outcomes in the intervention group will be compared to outcomes in the control group using multiple linear regression analysis, adjusting for possible confounders chosen prior to the analyses, i.e. sociodemographic variables.

In the economic evaluation study, a cost-utility analysis and a cost-effectiveness analysis will be performed from a societal perspective alongside the effectiveness study. The outcome in the cost-utility analysis will be quality-adjusted life years (QALYs) assessed by EQ-5D-5L measured at baseline and 12 months follow-up and valued by Danish preference weights. The outcome in the cost-effectiveness analysis will be changes in Mental Fatigue Scale. The costs of The Long COVID Rehabilitation Intervention will be estimated using micro-costing. Cost of usual rehabilitation will be estimated using micro-costing when possible or based on survey information from the municipalities. Visits to primary health care services will be extracted from the Danish National Health Service Register for Primary Care. Secondary healthcare services will be extracted from the National Patient Register. The valuation will be determined by the Diagnosis-Related-Grouping reimbursement rate and the outpatient-grouping-system. Productivity loss will be extracted from Danish Register for Evaluation of Marginalisation. The productivity costs per patient will be calculated using the Human Capital method.

To evaluate the cost-effectiveness of the intervention, the Incremental Cost-Effectiveness Ratio (ICER) will be calculated. Bias-corrected and accelerated bootstrapping with 10,000 replications will be performed to estimate 95% confidence intervals around cost differences and the uncertainty surrounding the ICERs. Uncertainty will be shown in cost-effectiveness plane. The cost-effectiveness acceptability curve will be drawn to show the probability that the intervention is cost-effective at different thresholds for willingness to pay for a gain in QALY or a clinical relevant improvement in Mental Fatigue Scale. Sensitivity analyses will be performed to test the robustness of the study results.

In the process evaluation study, the investigators will explore the processes of The Long COVID Rehabilitation Intervention by evaluating implementation, mechanism of impact and contextual factors. The study design is a concurrent mixed method study with quantitative and qualitative data collected and analysed during a similar timeframe. Implementation of the intervention will be investigated, focusing on fidelity, dose, adaptations and reach using patient baseline characteristics, routine monitored data from the patient' journals, and interviews with patients and health professionals. To evaluate mechanism of impact and contextual factors, the investigators will use a realist evaluation approach with pre-defined Context-Mechanism-Outcome configurations (CMOs) to explore under what circumstances, for whom, why and how the intervention works. This will be done using routine monitoring data from patient journals, individual interviews with patients (n=15) and focus group interviews with health professionals (n=5). An initial programme theory has been developed and graphically shown in a general logic model.

Quantitative and qualitative data are obtained and analysed simultaneously and linked at multiple points. Descriptive statistics will be used to analyse fidelity, dose and reach and will be presented with mean and standard deviation or median and percentiles as appropriate. Interview data will be transcribed verbatim and will be analysed following the standards for realist evaluations. The qualitative and quantitative results and most important CMOs will be merged to support refinement of the programme theory.

ELIGIBILITY:
Inclusion criteria:

* The patients should be diagnosed with long COVID and assessed at the Post-COVID-19 Clinic at Aarhus University
* The patients should be examined at the Department of Physiotherapy and Occupational Therapy and referred to rehabilitation in their municipality of residence
* The patients should be aged ≥ 18 years old
* The patients should be residing in one of the 19 municipalities of Central Denmark Region
* The patients should be referred to rehabilitation in their municipality of residence
* The patients should give informed written consent to participate in the study

Exclusion criteria:

* The patient is unable to give written informed consent (e.g. due to language barriers)
* The patient is resided outside of Central Denmark Region, Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long COVID examined at the Post-COVID-19 Clinic at Aarhus University Hospital and assessed at the Department of Physiotherapy and Occupational Therapy have been invited to participate in the project from July 2020 to June 2023. The patients are recruited to the study during their appointment at the Department of Physiotherapy and Occupational Therapy at Aarhus University Hospital for an examination of their functioning due to their long COVID symptoms. Thus, the inclusion of the patients is integrated into and carried out in clinical practise.
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The degree of mental fatigue measured with The Mental Fatigue Scale | At inclusion and 12-month follow-up
  The Mental Fatigue Scale measures the degree of mental fatigue through 15 questions covering affective, cognitive and sensory symptoms along with duration of sleep and daytime variation in symptom severity with a total score of 0-40. Higher score indicates higher degree of mental fatigue.
Number of weeks of sick leave obtained through the Danish Register for Evaluation of Marginalisation | From inclusion to 12-month follow-up
  The Danish Register for Evaluation of Marginalisation is a national register containing information on the Danish population. Sick leave is automatically registered when a person receives sick leave allowances.

SECONDARY OUTCOMES:
Health related quality of life estimated with the European Quality of Life - 5 Dimensions 5 Levels (EQ-5D-5L) | At inclusion and 12-month follow-up
  EQ-5D-5L is a self-assessed, health related, quality of life questionnaire measuring quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Disability estimated using The Post-COVID-19 Functional Status Scale | At inclusion and 12-month follow-up
  The Post-COVID-19 Functional Status Scale is an ordinal scale with six steps covering grade 0 (no functional limitations), grade 1 (negligible functional limitations), grade 2 (slight functional limitations), grade 3 (moderate functional limitations), grade 4 (severe functional limitations and grade 5 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Oestergaard Gregersen, PhD, Principal Investigator — DEFACTUM, Central Denmark Region, and Department of Public Health, Aarhus University
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark